CLINICAL TRIAL: NCT04254211
Title: Neutrophil-lymphocyte Ratio and Platelet-lymphocyte Ratio as Predictors for Adverse Events in Endovascular Aneurysm Repair for Abdominal Aorticaneurysm
Brief Title: Neutrophil-lymphocyte Ratio and Platelet-lymphocyte Ratio as Predictors for Adverse Events in EVAR
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: NLR, PLR in EVAR
Record Dates: First submitted 2020-01-05; First posted 2020-02-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Inflammation in EVAR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EVAR: Patinets with AAA, treated electively by EVAR. The values of simple inflammatory markers,neutrophil-lymphocyte ratio (NLR) and platelet-lymphocyte ratio (PLR), were measured pre- and postoperatively. Adverse events included any major adverse cardiovascular events (MACE), acute kidney injury and death from any cause
  Interventions: Other: NLR

INTERVENTIONS:
Other: NLR — neutrophil-lymphocyte ratio (NLR) and platelet-lymphocyte ratio (PLR)
  Other Names: PLR

SUMMARY:
This study investigated the association of chronic inflammatory markers with the clinical outcome after endovascular aneurysm repair (EVAR) for abdominal aortic aneurysm.

DETAILED DESCRIPTION:
The study included 230 consecutive AAA patients, treated electively by EVAR from March 2016 to February 2019. The values of simple inflammatory markers,neutrophil-lymphocyte ratio (NLR) and platelet-lymphocyte ratio (PLR), were measured pre- and postoperatively.Adverse events included any major adverse cardiovascular events (MACE), acute kidney injury and death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* AAA
* Elective
* EVAR

Exclusion Criteria:

* Emergency
* Open surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included consecutive AAA patients treated electively by EVAR
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
NLR major cardiovascular events (MACE) | Day 4 postopertively
  NLR indicator for major cardiovascular events (MACE)
PLR major cardiovascular events (MACE) | Day 4 postopertively
  PLR indicator for major cardiovascular events (MACE)
NLR acute kidney injury (AKI) | Day 4 postopertively
  NLR indicator for acute kidney injury (AKI)
PLR acute kidney injury (AKI) | Day 4 postopertively
  PLR indicator for acute kidney injury (AKI)
NLR death | Day 4 postopertively
  NLR indicator for death
PLR death | Day 4 postopertively
  PLR indicator for death

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly; Maria Ntalouka, MD, Principal Investigator — University Hospital of Larissa
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No